CLINICAL TRIAL: NCT06329453
Title: Intestinal Immunity in Neurologic Disease
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Erin E Longbrake, Principal Investigator, Yale University
Other Study IDs: 2000033081
Record Dates: First submitted 2024-01-29; First posted 2024-03-26 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis; Parkinson Disease; REM Sleep Behavior Disorder
MeSH Terms: conditions — Multiple Sclerosis; Parkinson Disease; REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Colon biopsies blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Individuals
  Interventions: Procedure: Colon Tissue Biopsy
- Individuals with neurologic diseases
  Interventions: Procedure: Colon Tissue Biopsy
- Individuals with known or suspected autoimmune diseases
  Interventions: Procedure: Colon Tissue Biopsy

INTERVENTIONS:
Procedure: Colon Tissue Biopsy — Colonoscopy and colon tissue biopsy.

SUMMARY:
The purpose of this study is to ascertain the functional profiles of the immune cells within the gastrointestinal tract and to determine how these cells contribute to autoimmune and neurologic diseases.

DETAILED DESCRIPTION:
Immune cells and microbes within the GI tract likely play an important role for neurologic disease pathogenesis, including MS and Parkinson's disease. Nevertheless, these immune cells have never been studied in detail using modern single cell technologies. Moreover, most of the human microbiome work done in this space to date has utilized fecal samples, but different anatomic niches within the gut may have greater importance for disease. This study will provide seminal information about how the relationships between gut immunity and neurologic/autoimmune diseases and may be paradigm shifting in regards to how the pathogenesis of some neurologic diseases is viewed.

This is an observational cohort study. Individuals undergoing colonoscopy (+/- upper endoscopy) as a part of standard of care or who consent to have a colonoscopy (+/- upper endoscopy) will be recruited to provide tissue biopsies obtained from the gastrointestinal mucosa. The rationale for including those who are not yet due to have a screening colonoscopy is that for many neurologic diseases (like MS), the disease onset is in adolescence or early adulthood, and the disease is diagnosed in young adults. These individuals would not yet be due to have screening colonoscopies, and yet changes in immune cells within the intestines may be a critical part of disease pathogenesis. This is what the investigators are exploring with this study.

The investigators will need to recruit age matched healthy controls because many features of the immune system change with age; as people get older, the immune system becomes less inflammatory ("immune senescence") and thus it is essential to have age-matched tissues for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and up

ONE of the following:

* Recommended to under a screening colonoscopy (+/- upper endoscopy) as part of standard of care. This includes healthy individuals as well as those with neurologic and/or autoimmune diseases. OR
* Willing to undergo research colonoscopy (+/- upper endoscopy) for research

Exclusion Criteria:

* Currently pregnant. Women of childbearing potential would perform a point of care urine pregnancy test prior to colonoscopy/endoscopy.
* Known or suspected, chronic inflammatory gastrointestinal disease (e.g. inflammatory bowel disease)
* Known, acute or chronic infections
* Systemic antibiotic (PO or IV) use within 3 months of colonoscopy
* Systemic corticosteroid use (equivalent of prednisone 10 mg per day or higher for >5 days) within 2 weeks of colonoscopy
* Malignancy, diagnosed or treated within the last 5 years
* Probiotic use within 2 weeks of procedure
* History of major GI surgery (e.g. colon resection, gastric bypass)
* Bleeding disorder, or on anticoagulant medication
* Other medical condition that, in the judgement of the investigator, would lead to higher-than-expected risks of biopsy
* Allergy to MAC anesthesia or other drugs used pursuant to standard of care for biospecimen collection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be individuals who are having screening colonoscopies (+/- upper endoscopies) and those who are willing to have these procedure/s performed for research, and who are willing to donate tissue for research. Healthy individuals, individuals with neurologic diseases, and individuals with known or suspected autoimmune diseases will all be candidates to participate
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Characterization of immune cells from the gastrointestinal mucosa | Through study completion, an average of 5 years
  Gastrointestinal mucosa cells will be characterized using sRNA measured through high-throughput sequencing with quantitative polymerase chain reaction (qPCR) validation.

SECONDARY OUTCOMES:
Evaluate spatial transcriptomics of intestinal tissue | Through study completion, an average of 5 years
  Spatial transcriptomics will be performed on gut mucosal biopsies
Characterize the microbiome at different anatomic sites within the gastrointestinal tract | Through study completion, an average of 5 years
  16S and/or shotgun metagenomic sequencing will be utilized to assess the composition of gut microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Erin Longbrake, Principal Investigator — Yale University
Locations (1):
- Yale MS Clinic, North Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No